CLINICAL TRIAL: NCT06199843
Title: Efficacy of Rifaximin vs Norfloxacin for Secondary Prophylaxis of SBP (NORRIF Trial): a Randomized Control Trial
Brief Title: Efficacy of Rifaximin vs Norfloxacin for Secondary Prophylaxis of SBP (NORRIF Trial)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-SBP-03
Record Dates: First submitted 2023-11-16; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-11

CONDITIONS: Spontaneous Bacterial Peritonitis
MeSH Terms: interventions — Rifaximin; Norfloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rifaximin (Experimental): Rifaximin 550 mg BD
  Interventions: Drug: Rifaximin
- Norfloxacin (Active Comparator): Norfloxacin 400 mg OD
  Interventions: Drug: Norfloxacin

INTERVENTIONS:
Drug: Rifaximin — Rifaximin 550 mg BD
  Arms: Rifaximin
Drug: Norfloxacin — Norfloxacin 400 mg OD
  Arms: Norfloxacin

SUMMARY:
SBP is a common complication of cirrhotics with associated increased mortality. After first episode of SBP there is increased risk of again developing SBP, with increased chance of developing resistant organism. So after the first episode of SBP, prophylaxis for prevention of second episode onwards is mandatory and therefore Rifaximin or Norfloxacin is considered. It has been seen that apart from preventing SBP they have other benefits with negligible side effects and therefore it is to be seen what other benefits including mortality benefits these drugs can confer.

DETAILED DESCRIPTION:
Hypothesis:-Rifaximin will be more effective in decreasing the incidence of SBP in patients with cirrhosis and prior episode of SBP

AIM:-.To study the efficacy and safety of Rifaximin vs Norfloxacin in preventing incident SBP, preventing non-SBP infections, and improving transplant free survival in patients with cirrhosis and previous episode of SBP

Methodology Single centered Open labeled Randomized Controlled Trial

Randomization will be done by block randomization method taking block size as 10. Data will be entered in Microsoft Excel and will be analysed by SPSS Version 28.Categorical Data will be represented as frequency (%) and will be analysed using Chi square or Fisher Exact Test as appropriate.Continuous Data will be represented as Mean +/- SD and compared using Student T test or Mann Whitney as per normality conditions are met or not.Beside this an appropriate analysis like survival analysis will be carried out at the time of Data Analysis.P value <0.05 will be considered as significant.

Rescue therapy: To be given to patients who develop SBP while on secondary prophylaxis, these patients will initially be treated by iv medication in hospital settings followed by change in therapy.

* Patients in Rifaximin limb developing SBP will switch to Norfloxacin
* Patients in Norfloxacin limb developing SBP will switch to Rifaximin

Treatment Failure: Defined as development of SBP at end of 6 months or 1 year of treatment.

Study population: age >18 years with prior incident SBP

Study design: Randomised case controlled trial

Study period: 1year after ethical clearance

Sample size: 280 (140 in each arm)

Intervention: This RCT will be conducted at ILBS New Delhi Monitoring and assessment: Monitoring will be done forall the parameters of the objective. Documentation will be done for any adverse effects which will happen.

STATISTICAL ANALYSIS: Assuming incidence of SBP over 6 months is 4% in Rifaximin & 15% in Norfloxacin Alpha 5% and power 80%. Enrollment of 260 cases (130 in each arm). Assuming dropout rate 10%.Total study cases calculated as 280 (140 in each arm). Random allocation in each arm by block method taking 10 as block size

ELIGIBILITY:
Inclusion Criteria:

1. Age>18 years
2. Cirrhosis (of any etiology) with ascites
3. Prior incident SBP

Exclusion Criteria:

1. Allergy to norfloxacin or rifaximin
2. Recent history of upper gastrointestinal bleed (UGIB) within 2 weeks
3. Patients with a history of multiple episodes of SBP
4. Patients with inoperable or not treatable HCC or other non-hepatic malignancy
5. Patients on immunosuppression
6. HIV infected
7. Post liver transplant
8. Recent (<6 months) abdominal surgery
9. Pregnant/lactating women
10. Other causes of ascites like tubercular or malignancy
11. Patients developing SBP on Norfloxcacin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-01-05 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of recurrence of SBP within 6 months | 6 months

SECONDARY OUTCOMES:
Incidence of recurrence of SBP within12 months | 12 months
Incidence of other site infections within 6 months | 6 months
Incidence of other site infections within 12 months | 12 months
to look for resistance pattern of infection in both norfloxacin and rifampicin group, type of resistant bacteria (MDR/XDR), and response of both groups to rifampicin and norfloxacin in secondary prophylaxis of SBP | 12 months
Incidence of other complications (HE, variceal bleed, Refractory ascites, AKI) within 6 months | 6 months
Incidence of other complications (HE, variceal bleed, Refractory ascites, AKI) within 12 months) | 12 months
Transplant free survival by 6 months | 6 months
Transplant free survival by 12 months | 12 months
Change in Child-Turcotte-Pugh (CTP) by 6 months | 6 months
Change in Model for End-Stage Liver Disease (MELD) scores by 6 months | 6 months
Change in Model for End-Stage Liver Disease Sodium (MELD Na) scores by 6 months | 6 months
Change in Child-Turcotte-Pugh (CTP) scores by 12 months | 12 months
Change in Model for End-Stage Liver Disease (MELD) scores by 12 months | 12 months
Change in MELD-Na scores by 12 months | 12 months
Side effects in both groups | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Jaya Benjamin, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided